CLINICAL TRIAL: NCT05726383
Title: MISTOSUS: Iscador® P (Mistletoe) Immunotherapy To Improve Event Free Survival In Patients With Relapsed Osteosarcoma After Resection Of Pulmonary Metastases
Brief Title: Iscador® P (Mistletoe) Immunotherapy for Recurrent Osteogenic Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Iscador AG, Arlesheim, Switzerland. (Unknown); Tackle Kids Cancer (Unknown); Susan Zabransky Hughes Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2021-1524
Record Dates: First submitted 2023-02-03; First posted 2023-02-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Osteogenic Sarcoma Recurrent
Keywords: Osteogenic; Sarcoma; Pulmonary; Metastatic; Immunotherapy; Mistletoe; Bone Tumor
MeSH Terms: conditions — Sarcoma; Neoplasm Metastasis; Bone Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm - Iscador*P (Experimental): Each Iscador® P therapy begins with a dose finding phase related to the drug' immunogenicity. In this phase, gradually increasing doses are used to determine the optimum individual dose response of the patient and to prevent excessive toxicity. The Iscador® P will be administered three times per week by subcutaneous injections (M,W,F) into the subcutaneous tissue of the thigh or abdomen. Treatment is administered according to a series of escalating doses that are given each of the three days in a week for 7 doses. There are 3 different series (Series 0, 1, and 2) and there are 7 dose vials in each series. Once the patient has reached their maximum tolerated dosing series, that series is used as the treatment regimen for the remaining weeks to a total duration of 52 weeks (13 cycles) or until disease progression. Each cycle is 4 weeks.
  Interventions: Drug: Iscador*P

INTERVENTIONS:
Drug: Iscador*P — Iscador P given for 2 cycles with follow up imaging done every 2 cycles. If imaging is negative patient remains on study for 13 cycles. If new lesion is found, then patient is off study.

SUMMARY:
This will be a phase II, single arm study of osteosarcoma patients with fully resected pulmonary metastases. The MTD corresponds to the dosage recommendations of the manufacturer of Iscador® P which is licensed in Sweden, New Zealand, South Korea, Germany and Switzerland for the treatment of solid tumors and precancerous lesions.

The study population includes patients with relapse of osteosarcoma in the lung following surgical resection of all gross disease (2nd or greater CR). Following completion of final thoracotomy, they will be treated with Iscador® P at concentrations up to the MTD with surveillance imaging via CT scan to monitor for relapsed disease.

DETAILED DESCRIPTION:
This will be a phase II, single arm study of osteosarcoma patients with fully resected pulmonary metastases. The MTD corresponds to the dosage recommendations of the manufacturer of Iscador® P which is licensed in Sweden, New Zealand, South Korea, Germany and Switzerland for the treatment of solid tumors and precancerous lesions.

Iscador® P is to be injected subcutaneously (abdominal) 3 times/week. All patients will start with Series 0 (0.01mg, 0.01mg, 0.1mg, 0.1mg, 1mg, 1mg, 1mg). If tolerated, they will receive this series for 2 consecutive boxes (2 x 7 vials per box). This will then be followed by Series 1 (0.1mg, 0.1mg, 1mg, 1mg, 10mg, 10mg, 10mg), which will be administered for the following 2 consecutive boxes (2 x 7 vials per box). If tolerated, patients will proceed to Series 2 (1mg, 1mg, 10mg, 10mg, 20mg, 20mg 20mg), which will be continued through week 52 (13 cycles).

The study population includes patients with relapse of osteosarcoma in the lung following surgical resection of all gross disease (2nd or greater CR). Following completion of final thoracotomy, they will be treated with Iscador® P at concentrations up to the MTD with surveillance imaging via CT scan to monitor for relapsed disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of osteosarcoma.
* Patients with at least one episode of relapse in the lung (without limitation of number of episodes), following surgical resection of all gross metastatic disease.
* Surgical resection of all possible sites of suspected pulmonary metastases in order to achieve a complete remission within 8 weeks prior to study enrollment. Note: If surgery related changes such as atelectasis are seen on the post-operative CT scan, patients will remain eligible to enroll as long as the operating surgeon believes that all sites of metastases were resected. Patients with positive microscopic margins will be eligible to enroll.
* Pathological confirmation of metastases from at least one of the resected sites.
* Age ≥ 8 years of age and <30 years of age.
* Patients must be able to receive subcutaneous injections.
* Performance level as measured by Karnofsky ≥60% for patients > 16 years of age or Lansky ≥ 60% for patients ≤ 16 years of age.
* Female patients of childbearing potential must have a negative serum blood pregnancy test during screening and a negative urine pregnancy test within 3 days prior to receiving the first dose of study drug. If the screening serum test is done within 3 days prior to receiving the first dose of study drug, a urine test is not required. If a patient is of childbearing potential the patient must agree to use effective contraception during the study and for 120 days after the last dose of study drug.
* If male, agrees to use an adequate method of contraception starting with the first dose of study drug through 120 days after the last dose of study drug
* Life expectancy of > two months
* Experienced resolution of toxic effect(s) of the most recent prior anti-cancer therapy to Grade <1 (except alopecia, cytopenia, or neuropathy). If a patient underwent major surgery or radiation therapy of >30 Gy, they must have recovered from the toxicity and/or complications from the intervention.
* Patients must meet the following laboratory criteria

  1. Adequate hepatic function with serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 times the upper limit of normal (ULN) and total serum bilirubin < 2.5 times the ULN or Direct bilirubin ≤ ULN for patients with total bilirubin levels > 2.5 X ULN
  2. Absolute neutrophil count ≥ 500/dL
  3. Platelet count ≥ 20,000/L
  4. Creatinine ≤ 1.5 X the ULN or measurement of calculated creatinine clearance (CrCl) ≥ 60 ml/minute

Exclusion Criteria:

* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator, including, but not limited to:

  * Another known malignancy other than osteosarcoma that is progressing or requires active treatment.
  * Any prior history of other cancer within the prior 5 years with the exception of adequately treated basal cell carcinoma or cervical intraepithelial neoplasia [CIN]/cervical carcinoma in situ or melanoma in situ).
  * Active infection requiring systemic therapy.
  * Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
  * New recurrence of osteosarcoma metastasis in any location other than lung
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study drug.
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Known active hepatitis B (e.g., hepatitis B surface antigen-reactive) or hepatitis C (e.g., hepatitis C virus ribonucleic acid [qualitative]). Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBc Ab] and absence of HBsAg) are eligible. HBV DNA test must be performed in these patients prior to study treatment. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Known history of chronic granulomatous diseases, florid autoimmune diseases, diseases treated with immunosuppressive drugs, hyperthyroidism with tachycardia, tuberculosis, parasitosis or Crohn's disease.
* If female, is pregnant or breastfeeding.
* Patients must have had no systemic chemotherapy or immunotherapy in the three weeks prior to enrollment and must have fully recovered from side effects of prior treatment at enrollment.
* Patients may not receive any additional chemotherapeutic agent (either conventional or experimental) while on study.
* Patients must not have received radiation therapy for up to two weeks prior to enrollment.
* Patients must have no known prior allergy to Iscador® P or any other Viscum album products.
* Patients must not receive concomitant treatment with immunostimulant or immunosuppressive drugs.

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2027-05-11 (Estimated); Study Completion 2027-05-11 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival | 12-months post complete resection of all metastases
  To estimate the event free survival for pediatric, adolescent and young adult patients with relapsed pulmonary osteosarcoma who are receiving treatment with subcutaneous Iscador® P following complete resection of all metastases.

SECONDARY OUTCOMES:
Quality of life post resection | 12-months post complete resection of all metastases
  Quality of life assessed with the NIH PROMIS® measures based on the patien's age. The PROMIS® Pediatric Profile v2.0 - Profile-25 and Parent-Proxy will be used for children from age 8 up to 18 years of age. It includes 25 questions with a graded categorical 5-point response scale.
  The PROMIS-29 Plus 2 Profile v2.1 for adults is a patient-reported measure of quality of life for adults. It includes 31 questions with a graded categorical 5-point response scale.
  Both PROMIS scales have a mean score of 50 and a standard deviation (SD) of 10 in the general population.
Time to relapse | 12-months post complete resection of all metastases
  Time to relapse in pediatric, adolescent, and young adult patients with relapsed pulmonary osteosarcoma who are receiving treatment with subcutaneous Iscador® P following complete resection of all metastases.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Offer, MD, Principal Investigator — Hackensack Meridian Health; Karen Moody, MD, Principal Investigator — MD Anderson
Locations (2):
- United States (2):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - M.D. Anderson Children's Cancer Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boye K, Longhi A, Guren T, Lorenz S, Naess S, Pierini M, Taksdal I, Lobmaier I, Cesari M, Paioli A, Londalen AM, Setola E, Hompland I, Meza-Zepeda LA, Sundby Hall K, Palmerini E. Pembrolizumab in advanced osteosarcoma: results of a single-arm, open-label, phase 2 trial. Cancer Immunol Immunother. 2021 Sep;70(9):2617-2624. doi: 10.1007/s00262-021-02876-w. Epub 2021 Feb 12. PMID 33580363
- [Background] Bussing A, Regnery A, Schweizer K. Effects of Viscum album L. on cyclophosphamide-treated peripheral blood mononuclear cells in vitro: sister chromatid exchanges and activation/proliferation marker expression. Cancer Lett. 1995 Aug 1;94(2):199-205. doi: 10.1016/0304-3835(95)03850-v. PMID 7634248
- [Background] Bussing A, Stumpf C, Troger W, Schietzel M. Course of mitogen-stimulated T lymphocytes in cancer patients treated with Viscum album extracts. Anticancer Res. 2007 Jul-Aug;27(4C):2903-10. PMID 17695469
- [Background] Chou AJ, Merola PR, Wexler LH, Gorlick RG, Vyas YM, Healey JH, LaQuaglia MP, Huvos AG, Meyers PA. Treatment of osteosarcoma at first recurrence after contemporary therapy: the Memorial Sloan-Kettering Cancer Center experience. Cancer. 2005 Nov 15;104(10):2214-21. doi: 10.1002/cncr.21417. PMID 16206297
- [Background] Gabius HJ, Gabius S, Joshi SS, Koch B, Schroeder M, Manzke WM, Westerhausen M. From ill-defined extracts to the immunomodulatory lectin: will there be a reason for oncological application of mistletoe? Planta Med. 1994 Feb;60(1):2-7. doi: 10.1055/s-2006-959396. PMID 8134410
- [Background] Gabriel AP, Mercado CP. Data retention after a patient withdraws consent in clinical trials. Open Access J Clin Trials. 2011 Apr;3:15-19. doi: 10.2147/OAJCT.S13960. PMID 23935390
- [Background] Horneber MA, Bueschel G, Huber R, Linde K, Rostock M. Mistletoe therapy in oncology. Cochrane Database Syst Rev. 2008 Apr 16;2008(2):CD003297. doi: 10.1002/14651858.CD003297.pub2. PMID 18425885
- [Background] Heinzerling L, von Baehr V, Liebenthal C, von Baehr R, Volk HD. Immunologic effector mechanisms of a standardized mistletoe extract on the function of human monocytes and lymphocytes in vitro, ex vivo, and in vivo. J Clin Immunol. 2006 Jul;26(4):347-59. doi: 10.1007/s10875-006-9023-5. Epub 2006 May 17. PMID 16705487
- [Background] Jung ML, Baudino S, Ribereau-Gayon G, Beck JP. Characterization of cytotoxic proteins from mistletoe (Viscum album L.). Cancer Lett. 1990 May 30;51(2):103-8. doi: 10.1016/0304-3835(90)90044-x. PMID 2344587
- [Background] Klein R, Classen K, Berg PA, Ludtke R, Werner M, Huber R. In vivo-induction of antibodies to mistletoe lectin-1 and viscotoxin by exposure to aqueous mistletoe extracts: a randomised double-blinded placebo controlled phase I study in healthy individuals. Eur J Med Res. 2002 Apr 30;7(4):155-63. PMID 12010650
- [Background] Klein R et al. Effects of mistletoe extracts on immunocompetent cells in vitro and in vivo and their relevance for the therapy of tumor diseases and other clinical entities. In Scheer R et al.(Ed): Forschritte in der Mistletherapie. KVC Verlag, Essen, 207-221. 2005
- [Background] Lagmay JP, Krailo MD, Dang H, Kim A, Hawkins DS, Beaty O 3rd, Widemann BC, Zwerdling T, Bomgaars L, Langevin AM, Grier HE, Weigel B, Blaney SM, Gorlick R, Janeway KA. Outcome of Patients With Recurrent Osteosarcoma Enrolled in Seven Phase II Trials Through Children's Cancer Group, Pediatric Oncology Group, and Children's Oncology Group: Learning From the Past to Move Forward. J Clin Oncol. 2016 Sep 1;34(25):3031-8. doi: 10.1200/JCO.2015.65.5381. Epub 2016 Jul 11. PMID 27400942
- [Background] Loef M, Walach H. Quality of life in cancer patients treated with mistletoe: a systematic review and meta-analysis. BMC Complement Med Ther. 2020 Jul 20;20(1):227. doi: 10.1186/s12906-020-03013-3. PMID 32690087
- [Background] Longhi A, Errani C, De Paolis M, Mercuri M, Bacci G. Primary bone osteosarcoma in the pediatric age: state of the art. Cancer Treat Rev. 2006 Oct;32(6):423-36. doi: 10.1016/j.ctrv.2006.05.005. Epub 2006 Jul 24. PMID 16860938
- [Background] Longhi A, Reif M, Mariani E, Ferrari S. A Randomized Study on Postrelapse Disease-Free Survival with Adjuvant Mistletoe versus Oral Etoposide in Osteosarcoma Patients. Evid Based Complement Alternat Med. 2014;2014:210198. doi: 10.1155/2014/210198. Epub 2014 Mar 31. PMID 24803944
- [Background] Longhi A, Cesari M, Serra M, Mariani E. Long-Term Follow-up of a Randomized Study of Oral Etoposide versus Viscum album Fermentatum Pini as Maintenance Therapy in Osteosarcoma Patients in Complete Surgical Remission after Second Relapse. Sarcoma. 2020 Apr 26;2020:8260730. doi: 10.1155/2020/8260730. eCollection 2020. PMID 32398946
- [Background] Meyers PA, Schwartz CL, Krailo MD, Healey JH, Bernstein ML, Betcher D, Ferguson WS, Gebhardt MC, Goorin AM, Harris M, Kleinerman E, Link MP, Nadel H, Nieder M, Siegal GP, Weiner MA, Wells RJ, Womer RB, Grier HE; Children's Oncology Group. Osteosarcoma: the addition of muramyl tripeptide to chemotherapy improves overall survival--a report from the Children's Oncology Group. J Clin Oncol. 2008 Feb 1;26(4):633-8. doi: 10.1200/JCO.2008.14.0095. PMID 18235123
- [Background] Olsnes S, Stirpe F, Sandvig K, Pihl A. Isolation and characterization of viscumin, a toxic lectin from Viscum album L. (mistletoe). J Biol Chem. 1982 Nov 25;257(22):13263-70. PMID 7142144
- [Background] Ostermann T, Appelbaum S, Poier D, Boehm K, Raak C, Bussing A. A Systematic Review and Meta-Analysis on the Survival of Cancer Patients Treated with a Fermented Viscum album L. Extract (Iscador): An Update of Findings. Complement Med Res. 2020;27(4):260-271. doi: 10.1159/000505202. Epub 2020 Jan 10. PMID 31927541
- [Background] Podlech O, Harter PN, Mittelbronn M, Poschel S, Naumann U. Fermented mistletoe extract as a multimodal antitumoral agent in gliomas. Evid Based Complement Alternat Med. 2012;2012:501796. doi: 10.1155/2012/501796. Epub 2012 Oct 22. PMID 23133496
- [Background] Schoffski P, Breidenbach I, Krauter J, Bolte O, Stadler M, Ganser A, Wilhelm-Ogunbiyi K, Lentzen H. Weekly 24 h infusion of aviscumine (rViscumin): a phase I study in patients with solid tumours. Eur J Cancer. 2005 Jul;41(10):1431-8. doi: 10.1016/j.ejca.2005.03.019. PMID 15913988
- [Background] Stammer RM, Kleinsimon S, Rolff J, Jager S, Eggert A, Seifert G, Delebinski CI. Synergistic Antitumour Properties of viscumTT in Alveolar Rhabdomyosarcoma. J Immunol Res. 2017;2017:4874280. doi: 10.1155/2017/4874280. Epub 2017 Jul 16. PMID 28791312
- [Background] Stein GM, Stettin A, Schultze J, Berg PA. Induction of anti-mistletoe lectin antibodies in relation to different mistletoe-extracts. Anticancer Drugs. 1997 Apr;8 Suppl 1:S57-9. doi: 10.1097/00001813-199704001-00013. PMID 9179370
- [Background] Stirpe F, Sandvig K, Olsnes S, Pihl A. Action of viscumin, a toxic lectin from mistletoe, on cells in culture. J Biol Chem. 1982 Nov 25;257(22):13271-7. PMID 7142145
- [Background] Timoshenko AV, Cherenkevich SN, Gabius HJ. Viscum album agglutinin-induced aggregation of blood cells and the lectin effects on neutrophil function. Biomed Pharmacother. 1995;49(3):153-8. doi: 10.1016/0753-3322(96)82609-6. PMID 7647287
- [Background] Twardziok M, Kleinsimon S, Rolff J, Jager S, Eggert A, Seifert G, Delebinski CI. Multiple Active Compounds from Viscum album L. Synergistically Converge to Promote Apoptosis in Ewing Sarcoma. PLoS One. 2016 Sep 2;11(9):e0159749. doi: 10.1371/journal.pone.0159749. eCollection 2016. PMID 27589063
- [Background] Wedekind MF, Wagner LM, Cripe TP. Immunotherapy for osteosarcoma: Where do we go from here? Pediatr Blood Cancer. 2018 Sep;65(9):e27227. doi: 10.1002/pbc.27227. Epub 2018 Jun 19. PMID 29923370
- [Background] Weissenstein U, Kunz M, Urech K, Regueiro U, Baumgartner S. Interaction of a standardized mistletoe (Viscum album) preparation with antitumor effects of Trastuzumab in vitro. BMC Complement Altern Med. 2016 Aug 4;16:271. doi: 10.1186/s12906-016-1246-2. PMID 27491866
- [Background] U.S. Department of Health and Human Services, Food and Drug Administration,Office of the Commissioner, Good Clinical Practice Program (2008). Guidance for Sponsors, Clinical Investigators, and IRBs Data Retention When Subjects Withdraw from FDA-Regulated Clinical Trials. From: https://www.fda.gov/media/75138/download. Accessed 7/22/20.
- [Background] Iscador AG, "ISCADOR in Cancer Therapy: Scientific Information and Study Results", www.iscador.com
- [Background] Iscador AG, "Iscador®P Investigational Medicinal Product Dossier (IMPD)" March, 2020 https://www.cancer.gov/about-cancer/treatment/cam/hp/mistletoe-pdq#_55. Accessed 12/30/19